CLINICAL TRIAL: NCT00046891
Title: The Use of Ginkgo Biloba For The Prevention Of Chemotherapy-Related Cognitive Dysfunction
Brief Title: EGb761 in Maintaining Mental Clarity in Women Receiving Chemotherapy for Newly Diagnosed Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N00C9; NCI-2012-02492 (Registry Identifier: CTRP (Clinical Trials Reporting System)); NCI-P02-0231; CDR0000257008 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Neurotoxicity
Keywords: neurotoxicity; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neurotoxicity Syndromes | interventions — Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginkgo Biloba (Experimental): 120 mg per day (60 mg BID)
  Interventions: Drug: Ginkgo Biloba
- Placebo (Placebo Comparator): 1 tablet BID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ginkgo Biloba — Patients will take 120 mg per day (60 mg BID)
  Arms: Ginkgo Biloba
Other: Placebo — Patients will take 1 tablet BID
  Arms: Placebo

SUMMARY:
RATIONALE: Chemotherapy may cause memory loss, attention loss, and other problems that make it difficult for patients to think clearly. EGb761 may help maintain mental clarity in patients undergoing chemotherapy.

PURPOSE: Randomized clinical trial to study the effectiveness of EGb761 in preventing loss of mental clarity in women who are receiving chemotherapy for newly diagnosed breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of EGb761 in the prevention of chemotherapy-related cognitive dysfunction in women with breast cancer.
* Determine the safety and tolerability of this drug when administered during adjuvant chemotherapy in these patients.
* Assess the onset and trajectory of cognitive loss that may occur during chemotherapy in these patients.
* Assess the quality of life and cognitive role functioning of patients treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to type of chemotherapy (doxorubicin/cyclophosphamide vs doxorubicin/cyclophosphamide with taxane vs other anthracycline-based chemotherapy vs other non-anthracycline-based chemotherapy), age (18 to 49 vs 50 and over), menopausal status at start of therapy (premenopausal vs postmenopausal vs unknown for surgical reasons), and lymph node involvement (0-3 vs 4 or more). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral EGb761 twice daily.
* Arm II: Patients receive oral placebo twice daily. Patients in both arms receive treatment beginning no later than the start of the second course of chemotherapy and continuing until 1 month after the completion of chemotherapy.

Quality of life and cognitive function are assessed at baseline, monthly during chemotherapy, and then at 1, 6, 12, 18, and 24 months.

Patients are followed every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 220 patients (110 per treatment arm) will be accrued for this study within 11 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed breast cancer
* Planned standard doses of adjuvant chemotherapy with or without a taxane

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Any status

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-1

Life expectancy

* At least 6 months

Hematopoietic

* No bleeding diathesis

Hepatic

* serum glutamate oxaloacetate transaminase (SGOT) no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 1.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No arterial vascular disease

Other

* Able to complete questionnaires alone or with assistance
* No diabetes
* No dementia
* No diagnosis of a psychiatric disorder within the past 5 years that would preclude study compliance
* No other significant comorbidity
* No known allergy to ginkgo biloba
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent stem cell transplantation

Chemotherapy

* No concurrent high-dose chemotherapy

Other

* More than 6 months since prior EGb761
* No concurrent antithrombotic therapy (e.g., daily aspirin or anticoagulants)

  * Anticoagulants used for central or peripheral line maintenance (i.e., warfarin 1 mg/day or heparin flushes) allowed
* No concurrent dose-intensive regimens
* No concurrent aspirin or aspirin-like medicines (e.g., indomethacin, ibuprofen, or some antihistamines or heparin or warfarin [except as used above])
* No concurrent regimen expected to cause thrombocytopenia
* No concurrent trazodone, monoamine oxidase inhibitors, or thiazide diuretics (e.g., chlorothiazide, hydrochlorothiazide, indapamide, or metolazone)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2002-12; Primary Completion 2006-10 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Study Chair — Mayo Clinic
Locations (175):
- United States (175):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Santa Barbara Hematology Oncology - Lompoc, Lompoc, California
  - Sansum Medical Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group at Cancer Center of Santa Barbara, Santa Barbara, California
  - Cancer Center of Santa Barbara, Snata Barbara, California
  - Santa Barbara Hematology Oncology - Solvang, Solvang, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Ochsner Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fergus Falls, Minnesota
  - Immanuel St. Joseph's Clinic, Mankato, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Sartell, Minnesota
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Hematology & Oncology Clinic, Hattiesburg, Mississippi
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Clinic of Dr. Judy L. Schmidt, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 226 patients were enrolled to this study between October 2002 and October 2006. There were 14 cancellations and 2 ineligible patients removed from the analysis; these participants were randomized but withdrew before beginning any study interventions. Efficacy analyses use all patients that reported baseline and one value after baseline.
Period: Overall Study
Arm/Group | Ginkgo Biloba | Placebo
Started | 113 | 113
Completed | 84 | 83
Not Completed | 29 | 30
Not completed — Cancels | 5 | 9
Not completed — Ineligible | 1 | 1
Not completed — Withdrawal by Subject | 18 | 15
Not completed — Adverse Event | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ginkgo Biloba | Placebo | Total
Number analyzed (Participants) | 113 | 113 | 226
Age, Customized [Number; unit: participants]
  Age < 50 | 55 | 54 | 109
  Age >= 50 | 58 | 59 | 117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 113 | 226
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 113 | 113 | 226

OUTCOME MEASURES:

1. Primary Outcome: The Level of Cognitive Dysfunction as Measured by the High Sensitivity Cognitive Screen (HSCS) Overall Score.
Description: The primary analysis involved compiling each subscale score for the HSCS into area under the curve (AUC) scores for the data points from baseline to the 12 month data point. HSCS instrument contains questions regarding Memory (0-39), Language (0-30), Visual-motor (0-10), Spatial (0-8), Attention and Concentration (0-25), Self-Regulation and Planning (0-6) on a varying scales. Total is calculated by summing afore mentioned subscales, values of Total ranged from 0 to 125. Lower scores are better.
Time Frame: Baseline, 12 months after starting Chemotherapy.
Population: Efficacy analyses uses all patients that reported baseline and one value after baseline.
Measure: Mean (Standard Deviation); unit: units on a scale*months
Arm/Group | Ginkgo Biloba | Placebo
Number analyzed (Participants) | 107 | 103
units on a scale*months
  Memory | 12.2 (9.18) | 12.6 (9.16)
  Language | 3.9 (6.84) | 2.6 (2.72)
  Visual-motor | 1.1 (1.29) | 0.7 (0.84)
  Spatial | 1.4 (0.92) | 1.3 (0.92)
  Attention/concentration | 2.2 (3.59) | 1.8 (2.16)
  Self-regulation | 2.4 (2.14) | 2.0 (2.10)
  Total | 20.7 (19.59) | 18.0 (12.26)
Statistical Analysis 1: Comparison: Ginkgo Biloba vs Placebo; Total HSCS Area Under the Curve (AUC) scores between the two treatment arms; Test type: Superiority or Other; p = 0.84, t-test, 2 sided

2. Secondary Outcome: Median Scores for Trail Making Tests A and B (Lower Scores Are Better).
Description: The Trail Making Test is a measure of overall brain dysfunction. Time taken to complete TMT tests was recorded. For this analysis median values of the Trail Making tests are calculated at different time points.
Time Frame: Baseline, 1, 6, 12, 18 and 24 months time points
Population: Secondary analyses uses all patients that reported data for all the time points.
Measure: Median (Full Range); unit: seconds
Arm/Group | Ginkgo Biloba | Placebo
Number analyzed (Participants) | 73 | 67
seconds
  TMT A: Baseline | 30 [15 to 270] | 28 [10 to 160]
  TMT A: 1 month | 25 [10 to 65] | 25 [8 to 65]
  TMT A: 6 months | 24 [10 to 48] | 22 [10 to 55]
  TMT A: 12 months | 23.5 [9 to 60] | 25 [12 to 75]
  TMT A: 18 months | 25 [10 to 75] | 23 [12 to 65]
  TMT A: 24 months | 23 [7 to 58] | 21 [10 to 50]
  TMT B: Baseline | 48 [20 to 417] | 50 [17 to 560]
  TMT B: 1 month | 45 [13 to 275] | 44 [20 to 100]
  TMT B: 6 months | 41 [20 to 99] | 42 [18 to 160]
  TMT B: 12 months | 40 [19 to 130] | 45 [18 to 180]
  TMT B: 18 months | 44.5 [10 to 145] | 40 [16 to 125]
  TMT B: 24 months | 40 [19 to 235] | 40 [19 to 143]

3. Secondary Outcome: Secondary Measure of Cognitive Function Using Trail Making Tests (TMT) A and B.
Description: TMT A and B were analyzed by evaluating median changes from baseline to different time points. Lower scores are better. The Trail Making Test will provide additional validity and verification for the assessment of overall cognitive dysfunction. Abbreviations used for category titles in the table below: Baseline (BL), change (chg), month (mth).
Time Frame: Baseline, 1, 6, 12, 18 and 24 months post chemotherapy.
Population: Secondary analysis uses all patients that reported baseline and at least one post baseline time point data.
Measure: Median (Full Range); unit: seconds
Groups:
- Ginko Bibola; Placebo: Median change from baseline to different time points.
Arm/Group | Ginko Bibola | Placebo
Number analyzed (Participants) | 107 | 103
seconds
  Chg in 1st Visit Post Chemo TMT A Score from BL | -4 [-237 to 20] | -4 [-117 to 21]
  Chg in 1st Visit Post Chemo TMT B Score from BL | -6.5 [-312 to 221] | -6.5 [-480 to 22]
  Chg in 6mth Visit Post Chemo TMT A Score from BL | -5 [-28 to 15] | -5 [-130 to 12]
  Chg in 6mth Visit Post Chemo TMT B Score from BL | -6.7 [-318 to 30] | -8 [-478 to 65]
  Chg in 12mth Visit Post Chemo TMT A Score from BL | -5 [-35 to 17] | -2 [-40 to 15]
  Chg in 12mth Visit Post Chemo TMT B Score from BL | -7 [-352 to 85] | -3 [-250 to 135]
  Chg in 18mth Visit Post Chemo TMT A Score from | -3.8 [-40 to 30] | -4 [-40 to 29]
  Chg in 18mth Visit Post Chemo TMT B Score from | -7 [-352 to 56.6] | -9 [-205 to 27]
  Chg in 24mth Visit Post Chemo TMT A Score from | -7 [-25 to 28] | -5 [-35 to 5]
  Chg in 24mth Visit Post Chemo TMT B Score from | -5 [-256 to 190] | -7 [-173 to 45]

4. Secondary Outcome: Self-reported Symptoms or Side Effects Using Symptom Experience Diary (SED)
Description: Self-reported symptoms or side effects mean change from baseline to 1st post chemo visit (negative numbers indicate worsening symptoms). A descriptive report of the toxicities experienced by participants will be measured with a Symptom Experience Diary. Participants will complete this questionnaire. This patient diary contains several questions related to potential side effects and side benefits of Ginko Biloba measured on a numeric analogue scale (based on 0-10 scale with 10 being worst toxicity).
Time Frame: Baseline, 1st evaluation of post chemotherapy.
Population: Secondary analyses uses all patients that reported data for baseline and post chemo visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginkgo Biloba | Placebo
Number analyzed (Participants) | 73 | 67
units on a scale
  Appetite loss | -0.5 (2.90) | -0.8 (2.81)
  Nausea | -0.1 (2.78) | -0.9 (2.67)
  Dizziness | -0.4 (1.96) | -0.3 (2.07)
  Constipation | -0.7 (2.77) | -0.9 (2.68)
  Headache | -0.6 (2.13) | -1.2 (2.31)
  Diarrhea | -0.3 (1.74) | 0.0 (2.10)
  Indigestion | 0 (2.61) | -0.4 (2.67)
  Bruising | -0.4 (2.33) | -0.9 (2.42)
  Overall QOL | -0.4 (2.08) | -0.6 (2.40)
  Thinks memory affects QOL | 0.5 (2.82) | -0.5 (3.06)

5. Secondary Outcome: Associations Between Self-reported Cognition and the HSCS.
Description: Pearson correlation coefficients conceptually related objective HSCS and subjective self-reported cognition. For this analysis data from both arms are combined. In the table below, numbers closer to 1 indicate positive correlation; numbers closer to -1 indicate negative correlation.
Time Frame: Baseline, 1, 6, 12, 18 and 24 months time points
Population: Secondary analyses uses all patients that reported data for baseline and one of the post baseline time points.
Measure: Number; unit: Pearson correlation coefficient
Groups:
- Stay Focused; Think Clearly; Balance Checkbook: Self-report cognition
Arm/Group | Stay Focused | Think Clearly | Balance Checkbook
Number analyzed (Participants) | 158 | 158 | 158
Pearson correlation coefficient
  HSCS attention concentration at 1 month | 0.01 | 0.08 | -0.02
  HSCS attention concentration at 6 months | -0.06 | 0.00 | -0.02
  HSCS attention concentration at 12 months | -0.02 | 0.02 | -0.08
  HSCS attention concentration at 18 months | 0.14 | 0.07 | -0.10
  HSCS attention concentration at 24 months | -0.06 | -0.07 | -0.10

6. Secondary Outcome: Associations Between Self-report Measures of Cognition and the Trail Making Test (TMT) A and B.
Description: Pearson correlation coefficients conceptually related objective TMT A and B and subjective self-report measures of cognition. For this analysis data from both arms are combined. In the table below, numbers closer to 1 indicate positive correlation; numbers closer to -1 indicate negative correlation.
Time Frame: Baseline, 1, 6, 12, 18 and 24 months time points
Population: Secondary analyses uses all patients that reported data for baseline and one of the post baseline time points.
Measure: Number; unit: Pearson correlation coefficient
Groups:
- Solve Problems; Plan Ahead; Make Decisions: Self-report cognition
Arm/Group | Solve Problems | Plan Ahead | Make Decisions
Number analyzed (Participants) | 158 | 158 | 158
Pearson correlation coefficient
  TMT A at 1 month | -0.01 | 0.05 | -0.05
  TMT A at 6 months | 0.04 | .20 | 0.10
  TMT A at 12 months | -0.09 | 0.03 | -0.01
  TMT A at 18 months | 0.06 | 0.08 | 0.08
  TMT A at 24 months | -0.01 | -0.02 | -0.02
  TMT B at 1 month | -0.08 | -0.02 | -0.06
  TMT B at 6 months | 0.09 | 0.28 | 0.21
  TMT B at 12 months | 0.13 | 0.16 | 0.10
  TMT B at 18 months | 0.06 | 0.08 | 0.10
  TMT B at 24 months | 0.00 | -.05 | 0.00

ADVERSE EVENTS:
Time Frame: 12 months during treatment.
Description: Total of 104 and 101 patients from Ginko and placebo arms respectively are evaluable for toxicity evaluation. There were 14 cancellations and 2 ineligible patients removed from the analysis. Five patients went off study before they were evaluated for toxicity.
Arm/Group | Ginkgo Biloba | Placebo
Serious Adverse Events (participants affected / at risk) | 4/104 | 3/101
Other Adverse Events (participants affected / at risk) | 89/104 | 94/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ginkgo Biloba (N=104) | Placebo (N=101)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (6) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ginkgo Biloba (N=104) | Placebo (N=101)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 66 (186) | 72 (186)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis due to radiation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 68 (151) | 66 (159)
Vomiting (Gastrointestinal disorders) | 32 (53) | 37 (64)
Chest pain (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 6 (6) | 5 (6)
Pain (General disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 2 (2) | 2 (2)
Wound-infectious (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 56 (119) | 60 (126)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 15 (21) | 13 (20)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 25 (58) | 32 (53)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hemorrhage (Vascular disorders) | 19 (26) | 17 (25)
Thrombosis (Vascular disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes